CLINICAL TRIAL: NCT06434805
Title: An Education Initiative to Reduce Stigma Towards Sex Workers and Sexual Minorities Among Nursing Students: a Pilot Study
Brief Title: An Education Initiative to Reduce Stigma Towards Sex Workers and Sexual Minorities Among Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Polly MA Haixia, Assistant Professor, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HE-NHS2024/02
Record Dates: First submitted 2024-05-18; First posted 2024-05-30 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-11

CONDITIONS: Stigmatization; Sex Work; Homosexuality; Transgenderism
Keywords: gender and sexual minority; sex workers; cultural competency; nursing students
MeSH Terms: conditions — Stereotyping; Sex Work; Homosexuality; Transsexualism; Coitus

STUDY DESIGN:
Intervention Model Description: A single group with outcome assessments will be taken at baseline, immediately after the intervention, and at 2-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Education workshop (Other): This is a one-day workshop with four sessions.
  Interventions: Other: sex workers and sexual minorities education workshop

INTERVENTIONS:
Other: sex workers and sexual minorities education workshop — The participants will receive a one-day workshop (four sessions). The generic content aims at enhancing the understanding of sexual orientation, gender identities, social stigma, sex work and sexual orientation and human rights (session 1), the lived experience of SWSM (session 2), the content specifically related to the medical and healthcare field, including be familiar with the professional and ethical obligations (session 3), the skills that can be adopted when providing services to SWSM (session 4).

SUMMARY:
Background: Sex workers and sexual minorities (SWSM) often encounter barriers when accessing healthcare services due to social stigma and discrimination. In Hong Kong, stigma and prejudice exist among nurses and nursing students toward SWSM.

Aims: This education initiative aims to improve the knowledge, attitudes, and clinical competence of nursing students in caring for SWSM.

Methods: This pilot study will employ a one-group pre-and post-test design. Convenience sampling will be used to recruit 32 nursing students from the clinical phase of the Bachelor of Nursing program at the School of Nursing and Health Studies of Hong Kong Metropolitan University, as well as nursing students from other local universities. The intervention will consist of a four-session one-day workshop based on social cognitive theory and interpersonal contact theory. The workshop will cover various topics, including terminologies, human rights, stigma and discrimination in healthcare settings, contact with SWSM, and skills building. The primary outcome measure will include participants' attitudes toward SWSM. Secondary outcome measures included their knowledge and clinical competence. These outcome measurements will be assessed at baseline (T0) and immediately after the intervention (T1) and two months follow up (T2). Additionally, focus group discussions will be carried out to explore participants' experiences of the intervention.

Discussion: Findings from this study could contribute to the existing knowledge on stigma surrounding SWSM in Hong Kong and its impact on healthcare. The intervention is expected to increase the knowledge, attitudes, and skills of nursing students in providing care for SWSM. By promoting non-judgmental and equitable care, the research aims to contribute to the overall well-being and health outcomes of SWSM. These results will inform future nursing education curricula and clinical practice, facilitating the development of more inclusive and patient-centered care for marginalized populations in Hong Kong and beyond.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years of age or above;
* studying in the clinical phase (i.e., year 3 to year 5);
* are able to speak, read, and write Cantonese or Putonghua;
* are willing to participate in the study and share their experience of the education initiative with the research group;
* have informed consent to participate in the study.

Exclusion Criteria:

* Those who have completed a similar workshop or discussion of sex workers and sexual minorities in previous nursing education will be excluded from this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
LGBT development of clinical skills scale (LGBT-DOCSS) | baseline, immediately after the intervention, 2-months post-intervention
  LGBT-DOCSS will be used to assess nursing students' clinical skills in caring for sexual minorities. It includes 18 items crossing three domains: clinical preparedness, attitudinal attitudes, and basic knowledge. A 7-point Likert-type scale was used, with 1 = not at all true, 4 = somewhat true, and 7 = total true. The total score ranges from 18 to 126. Higher scores are indicative of higher levels of clinical preparedness and rudimentary knowledge and less prejudicial attitudinal awareness regarding LGBT clients/patients. LGBT-DOCSS was back-and-forth translated by the research team.

SECONDARY OUTCOMES:
Acceptability of the workshop | baseline, immediately after the intervention, and 2-month follow-up.
  Participants' acceptability of the workshop was assessed using self-developed questionnaire consisting 10 items. Each item was rated on a five-point Likert scale (1 = strongly disagree, 5 = strongly agree). Example of the items included evaluations of the appropriateness, relevance, diversity, and interest of the content, and participants' confidence in caring for LGBTQ+ people after the workshop, their overall satisfaction with the experience, and their willingness to recommend it to others.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Participants' privacy, confidentiality, and voluntary participation of the study will be ensured. Participants' information will be kept in a password-protected computer. Only the research team could access the original data.